CLINICAL TRIAL: NCT05738109
Title: Evaluating the Efficacy of a 91-day Self-talk Mental Health Self-care Journal
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Victoria (Other)
Collaborators: Switch Research (Unknown); Mathematics of Information Technology and Complex Systems (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 21-0361
Record Dates: First submitted 2023-02-03; First posted 2023-02-21 (Actual); Last update posted 2024-06-14 (Actual); Status verified 2023-12

CONDITIONS: Mental Health; Self Care
Keywords: mental health; self-care; self-talk; pilot trial
MeSH Terms: conditions — Psychological Well-Being

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Self-guided journaling Intervention (Experimental): Participants assigned to the waitlist group complete a 2wk, 1mo, 2mo and 3mo survey over the 91-day study period. After the 91-days they will also complete a follow-up survey and exit interview
  Interventions: Other: Self-Talk Journals
- Waitlist Control (No Intervention): Participants assigned to the waitlist group complete a 2wk, 1mo, 2mo and 3mo survey over the 91-day study period. After the 91-days they receive access to the 91-day Self-Talk Journal for their own personal use.

INTERVENTIONS:
Other: Self-Talk Journals — Participants randomized to the intervention group will receive a physical copy of the 91-day self-talk journal during the baseline meeting. Participants will also be introduced the purpose of the journal and its intended usage (i.e., daily journaling). Intervention participants will not be offered guidance or feedback on the journal after these initial instructions, in order to emulate an ad libitum usage. Control group participants will not receive any contact with the researchers outside of the planned questionnaires and to receive their journal at the three-month timepoint.
  Arms: Self-guided journaling Intervention

SUMMARY:
1. Does a 91-day self-talk journal intervention improve outcomes of self-criticism, self-esteem, automatic negative self-statements, and mental health among participants using the journal over wait-list control?
2. What is the adherence rate to a 91-day self-talk journal intervention?
3. What were participants' experience(s) of using a 91-day self-talk journal?

DETAILED DESCRIPTION:
The following research project can contribute to the investigators' understanding of how/how well self-guided resources can increase participant outcomes of self-criticism, self-esteem, automatic negative self-statements, and mental health. Self-guided resources such as a self-talk journal provide can provide an easily accessible avenue for improving individual mental health. There has been a recent surge in the popularity of health-promotive self-care products, or products aimed at providing individuals with "the knowledge, skills, and attitudes required to achieve and maintain good health". These products (often in the form of journals) are similar to "self-help books"; however, a key difference is that self-care products prompt and provide space for the reader to actively engage in activities and psychological techniques, unlike the passive nature of traditional self-help books. These products typically address mental health concerns (i.e., mental health self-care) and are advertised to provide an effective means for individuals to reduce stress, improve self-compassion, and boost wellbeing. What's more, the generally positive reviews these products garner provides the perception that these products are well-received and effective in eliciting these outcomes. However, the scientific foundation for the majority of these journals is unknown. Furthermore, the efficacy of these products for improving or promoting their intended outcome(s) is often not addressed outside of these, often positive, reviews.

ELIGIBILITY:
Inclusion Criteria:

(1) being 19+ years old, (2) being fluent in English, (3) currently living in the Greater Victoria area, (4) self-reporting no previously diagnosed mental illness or psychiatric conditions, and (5) scoring >12 on the Self-Criticism subscale of the Self-Talk Scale (based on previous mean data; Brinthaupt, Hein, & Kramer, 2009).

Exclusion Criteria:

* Scoring =<12 on the Self-Talk Scale, currently receiving or seeking therapy for a mental illness, or a current or previous diagnosis of mental illness.

Min Age: 19 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 67 (Actual)
Dates: Start 2022-09-13 (Actual); Primary Completion 2024-04-30 (Actual); Study Completion 2024-04-30 (Actual)

PRIMARY OUTCOMES:
Self-Talk. | Change from baseline at 2 weeks, 1 month , 2 months, and 3 months for all participants. As well as 4 months for intervention participants
  Assessed using the Self-Talk Scale. The scale consists of 16 items rated on a five-point frequency scale (1 = never, 5 = very often) using the common stem "I talk to myself when…"
  It has a four factor-structure comprised of self-assessment, self-reinforcement, self-criticism and self-management.
  Total scores range from 16-80. Individual subscales scores range from 16-20. The higher the score the greater frequency of one's self-talk.

SECONDARY OUTCOMES:
Self-esteem | Change from baseline at 2 weeks, 1 month , 2 months, and 3 months for all participants. As well as 4 months for intervention participants
  Assessed using the Rosenberg Self-Esteem Scale, a 10-item measure of global self-esteem or self-worth.
  Uses a 4-point likert scale ranging from 1 (strongly agree) to 4 (strongly disagree)
  Possible scores range from 10-40, higher scores indicate higher levels of self-esteem
Self-consciousness | Change from baseline at 2 weeks, 1 month , 2 months, and 3 months for all participants. As well as 4 months for intervention participants
  Aspects of self-consciousness, including private self-consciousness, internal state awareness, self-reflection, public self-consciousness, and social anxiety, will be assessed using the Fenigstein Self-Consciousness Scale.
  The scale consists of 23 items, rated using a 5-point likert scale ranging from 0 (extremely uncharacteristic) to 4 (extremely characteristic), with higher scores denoting higher levels of self-consciousness.
Automatic Negative Self-Statements | Change from baseline at 2 weeks, 1 month , 2 months, and 3 months for all participants. As well as 4 months for intervention participants
  The frequency of automatic negative self-statements will be assessed using the Automatic Thoughts Questionnaire, whose 30-items assess the frequency of negative self-statements associated with depression.
  Uses a 5-point likert scale comprised of the following: 1 = not at all, 2 = sometimes, 3 = moderately often, 4 = often , and 5 = all of the time. Possible scores range from 30-150, with higher scores indicating greater rates of negative self-statements.
Adherence to Journal | Change from baseline at 2 weeks, 1 month , 2 months, and 3 months for all participants. As well as 4 months for intervention participants
  Adherence to the journal for the intervention group will be assessed using three items:
  1. "Currently, what is the last day of the journal [the participant] completed?": possible score range 0-91, 0 indicates no days have been completed
  2. "[Has the participant] skipped or not completed any days prior to the latest day [the participant] completed?": No or yes - indicate which days
  3. "Approximately how many minutes [did the participant] spend completing a day, within the journal?": self-reported number of daily minutes
Experience using the journal. | At 3 months from baseline or if and when intervention participants drop out of the study
  Intervention group participants' experience using the journal will be assessed through a qualitative exit interview
Demographics | Baseline
  Age, preferred gender, socio-economic status, ethnicity, educational attainment, and employment status will be collected
Mental Health | Change from baseline at 2 weeks, 1 month , 2 months, and 3 months for all participants. As well as 4 months for intervention participants
  Depression and anxiety will be assessed using the Hospital Anxiety and Depression Scale.
  Possible scores for each subscale range from 0-21. A score of 0-7 = "normal", 8-10 = "Borderline abnormal (borderline case)" and 11-21 = "Abnormal (case)."
Subjective Well-Being | Change from baseline at 2 weeks, 1 month , 2 months, and 3 months for all participants. As well as 4 months for intervention participants
  Subjective well-being will be assessed using the Warwick-Edinburgh Mental Wellbeing Scale.
  Uses a 5-point Likert scale: 1= none of the time, 2= rarely, 3 = some of the time, 4 = often, and 5 = all of the time. Possible scores range from 14 to 70, with higher scores indicating greater mental-wellbeing
Physical Activity, Sedentary Behaviour and Sleep | Change from baseline at 2 weeks, 1 month , 2 months, and 3 months for all participants. As well as 4 months for intervention participants
  Modified International Physical Activity Questionnaire includes open-ended questions surrounding individuals':
  1. Physical activity. Frequency score ranging from 0-7 days per week. Average time spent on one of those days ranging from 0-24 total hours. Separate questions for vigorous intensity, moderate intensity, mild intensity and walking.
  2. Sitting reported in average hours per day ranging from 0-24 total hours.
  3. Occupational and recreational screentime. Reported using a separate daily average for weekdays and weekends ranging from 0-24 total hours.
  4. Sleep reported using average number of hours per night ranging from 0-24 total hours.

CONTACTS AND LOCATIONS:
Overall Officials: Ryan Rhodes, PhD, Principal Investigator — Lab Director and Professor
Locations (1):
- Behavioural Medicine Lab UVic, Victoria, British Columbia, Canada

IPD SHARING:
Plan to Share IPD: No